CLINICAL TRIAL: NCT02789657
Title: Efficacy of Carboplatin and Paclitaxel With Trastuzumab and Pertuzumab (wPCbTP) and Switching to an Anthracycline-based Regimen (AC) in Non-responding Patients in Clinical Stage I-III HER2-positive Breast Cancer.
Brief Title: Neoadjuvant Therapy in Clinical Stage I-III HER2-positive Breast Cancer.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Brown University (Other)
Collaborators: Women and Infants Hospital of Rhode Island (Other); Rhode Island Hospital (Other); The Miriam Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BrUOG 308
Record Dates: First submitted 2016-05-30; First posted 2016-06-03 (Estimated); Results first posted 2022-04-28 (Actual); Last update posted 2022-05-19 (Actual); Status verified 2022-04

CONDITIONS: Breast Cancer
Keywords: neoadjuvant breast cancer; stage I-III breast cancer; HER 2 positive breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Paclitaxel; Trastuzumab; pertuzumab; Carboplatin; Mastectomy, Segmental

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Optimal- 18 weeks (Experimental): 18 weeks (6 cycles) of paclitaxel, carboplatin, trastuzumab and pertuzumab. Post treatment, patients will undergo surgery.
  Interventions: Drug: paclitaxel; Drug: Trastuzumab; Drug: Pertuzumab; Drug: carboplatin; Procedure: Breast surgery
- Sub-optimal with AC (Experimental): 12 weeks (4 cycles) of paclitaxel, carboplatin, trastuzumab and pertuzumab. Post 12 weeks, initiation of doxorubicin and cyclophosphamide for 4 cycles (6 weeks), followed by surgery.
  Interventions: Drug: paclitaxel; Drug: Trastuzumab; Drug: Pertuzumab; Drug: carboplatin; Procedure: Breast surgery; Drug: AC
- Optimal with AC (Experimental): Less than 18 weeks (6 cycles) of paclitaxel, carboplatin, trastuzumab and pertuzumab, followed by initiation of doxorubicin and cyclophosphamide. Post treatment, patients will undergo surgery.
  Interventions: Drug: paclitaxel; Drug: Trastuzumab; Drug: Pertuzumab; Drug: carboplatin; Procedure: Breast surgery; Drug: AC
- Sub-optimal no AC (Experimental): 18 weeks (6 cycles) of paclitaxel, carboplatin, trastuzumab and pertuzumab. Post treatment, patients will undergo surgery.
  Interventions: Drug: paclitaxel; Drug: Trastuzumab; Drug: Pertuzumab; Drug: carboplatin; Procedure: Breast surgery

INTERVENTIONS:
Drug: paclitaxel — 80 mg/m2 (or nab-paclitaxel 80-100 mg/m2) weekly
  Other Names: taxel, onxal
Drug: Trastuzumab — Either every 3 weeks (8 mg/kg cycle 1 then 6 mg/kg cycles 2-4) or weekly (4 mg/kg week 1 then 2 mg/kg weeks 2-12)
  Other Names: Herceptin
Drug: Pertuzumab — every 3 weeks (840 mg cycle 1 then 420 mg cycles 2-4) or weeks 1 and 2 cycle 1 (420 mg each dose) during the first 3-6 weeks of treatment, then 420 mg day 1 of cycles 2-4.
  Other Names: Perjeta
Drug: carboplatin — AUC 2 administered weekly with no planned treatment breaks
  Other Names: paraplatin
Procedure: Breast surgery — breast conserving or mastectomy
Drug: AC — doxorubicin and cyclophosphamide (AC) every 2 or 3 weeks for 4 cycles
  Dose-dense AC: Doxorubicin 60 mg/m2 and cyclophosphamide 600 mg/m2 IV day 1 every 2 weeks x 4 cycles
  Standard AC: Doxorubicin 60 mg/m2 and cyclophosphamide 600 mg/m2 IV day 1 r every 3 weeks x 4 cycles
  Arms: Optimal with AC; Sub-optimal with AC

SUMMARY:
Neoadjuvant therapy is given to breast cancer patients whose cancers are relatively large or have spread to lymph nodes or both. The primary goal of this treatment is to prevent the cancer from coming back (recurring) elsewhere in the body, but if it makes the cancer in the breast and lymph nodes shrink it might be easier to remove. This could allow a patient to have a lumpectomy instead of a mastectomy and reduce the number of lymph nodes that the surgeon has to remove. In some cases, the neoadjuvant therapy works so well that it kills all of the cancer in the breast and lymph nodes. This is referred to as a pathologic complete response (pCR). Patients who achieve a pCR have a much lower risk of the cancer recurring elsewhere in their bodies.

Investigators aren't sure which chemotherapy drugs work best with the HER2-targeted drugs, and what combination of these drugs causes the fewest side effects.Thus, this study has two main goals:

1. To find out if treatment with wPCbTP, weekly paclitaxel and carboplatin given with trastuzumab and pertuzumab every 3 weeks, leads to as many pCRs as TCHP in patients with HER2-positive breast cancer, but has fewer side effects.
2. To find out if HER2-positive patients whose cancers are not responding well after 12 weeks of wPCbTP get a better response when they are switched to a doxorubicin-containing regimen called AC for 4 cycles (8-12 weeks).

DETAILED DESCRIPTION:
See summary above

ELIGIBILITY:
Inclusion Criteria:

1 Histologically confirmed adenocarcinoma of the breast, with sufficient tissue available from needle or incisional biopsy (excisional biopsy not permitted) for ER, PR and HER2 testing.

2. Resectable - clinical stage I (only with T=2.0 cm), IIA-IIIA - T2 N0-T3N0 or T1-3 N1-N2a - or unresectable - clinical stage IIIB-C - T4 or N2b-3 - disease. No evidence of M1 disease. Pretreatment clinical stage will be recorded by the treating physician.

3. Breast tumor measuring at least 1 cm in greatest dimension by ultrasound or MRI; patients without measurable disease in the breast (TX) by imaging studies are eligible if they have measurable disease (a node measuring at least 1 cm along its short axis, and histologically confirmed to contain metastatic disease) in the axilla.

4. HER2+, defined by either IHC 3+ or amplification of the HER2 gene by FISH analysis (ratio >2.0 or >6 HER2 targets per cell; patients with equivocal HER2 testing, 2+ by IHC with a FISH ratio of <2.0 and 4-6 HER2 signals per nucleus, are not eligible).

5. Patients with multiple foci of invasive cancer in the same breast are eligible if any single lesion meets the above size criteria and all sampled lesions > 1 cm in maximum dimension are histologically similar and HER2+. Patients are also eligible , or if there is a focus of HER2- invasive cancer that is <1 cm in maximum dimension and in a different quadrant of the breast from the HER2+ cancer, such that its presence will not interfere with clinical or pathologic assessment of response of the HER2+ cancer. The presence of DCIS or LCIS in either breast will not render a patient ineligible. Patients with a small focus of invasive cancer detected in the contralateral breast (clinical T1a/bN0) are eligible, whether the contralateral tumor is HER2+ or HER2-, while patients with a more advanced invasive cancer in the contralateral breast are not eligible; in patients with a small focus of invasive cancer in the contralateral breast or a small focus of HER2- cancer in the same breast only the histologic response in the HER2+ target lesion will be considered in determining the patient's pathologic response.

6 It is recommended that patients have a pretreatment echocardiogram or MUGA scan with an LVEF above the institutional lower limit of normal.

7. Female, age >18, Zubrod PS 0-1. 8. It is recommended that patients have adequate bone marrow, renal and hepatic function. Examples of this include: ANC > 1000/ul, platelet count >100,000/ul, HGB> 9.0 g/dl, serum creatinine <1.5 mg/dl or measured creatinine clearance of >30 ml/min and AST <5 x ULN.

9. Signed informed consent.

Exclusion Criteria:

1. Prior chemotherapy, hormonal therapy, or radiation therapy for this cancer
2. Patients with congestive heart failure, unstable angina pectoris, absolute exclusion for BP >180 (systolic) or >100 (diastolic); for BP 160-180/90-100, assurance from the treating MD that this is being addressed and that the MD is comfortable initiating study treatment despite the elevated value(s)uncontrolled clinically significant arrhythmia or grade II or greater peripheral vascular disease are not eligible. Patients with BP >180 (systolic) or >100 (diastolic) are excluded; patients with BP 160-180/90-100 are eligible with assurance from the treating MD that this is being addressed and that the MD is comfortable initiating study treatment despite the elevated value(s).
3. Patients with myocardial infarction, stroke or arterial thrombotic event within the past 12 months are not eligible.
4. Pregnant and lactating women are not eligible. All patients of reproductive potential should have a negative pregnancy test at baseline and be advised to use an effective barrier method of contraception if sexually active during treatment on the study and for 2 months post the last treatment. Sites will be asked to confirm the patient's menopausal status at study entry and that premenopausal women had a negative pregnancy test performed within 7 days of starting treatment, but will not be required to submit test results.
5. Active (defined as symptomatic, currently requiring treatment or likely to require treatment within the 6 months following study enrollment, or likely to affect the efficacy or tolerability of the study treatment) non-breast malignancy.
6. Baseline grade >2 peripheral neuropathy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2016-11-21 (Actual); Primary Completion 2019-11-14 (Actual); Study Completion 2020-03-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Howard Safran, MD, Study Chair — BrUOG Study Chair
Locations (2):
- United States (2):
  - Rhode Island Hospital and The Miriam Hospital, Providence, Rhode Island
  - Women and Infants hospital of RI, Providence, Rhode Island

REFERENCES:
- [Derived] Lopresti ML, Bian JJ, Sakr BJ, Strenger RS, Legare RD, Fenton M, Witherby SM, Dizon DS, Pandya SV, Stuckey AR, Edmondson DA, Gass JS, Emmick CM, Graves TA, Cutitar M, Olszewski AJ, Sikov WM. Neoadjuvant weekly paclitaxel and carboplatin with trastuzumab and pertuzumab in HER2-positive breast cancer: a Brown University Oncology Research Group (BrUOG) study. Breast Cancer Res Treat. 2021 Aug;189(1):93-101. doi: 10.1007/s10549-021-06266-9. Epub 2021 Jun 4. PMID 34086171

RESULTS

PARTICIPANT FLOW:
Groups:
- Experimental: Optimal- 18 Weeks; Experimental: Sub-optimal no AC: 18 weeks (6 cycles) of paclitaxel, carboplatin, trastuzumab and pertuzumab. Post treatment, patients will undergo surgery.
- Experimental: Sub-optimal With AC: 12 weeks (4 cycles) of paclitaxel, carboplatin, trastuzumab and pertuzumab. Post 12 weeks, initiation of doxorubicin and cyclophosphamide for 4 cycles (6 weeks), followed by surgery.
- Experimental: Optimal With AC: Less than 18 weeks (6 cycles) of paclitaxel, carboplatin, trastuzumab and pertuzumab, followed by initiation of doxorubicin and cyclophosphamide. Post treatment, patients will undergo surgery.
Period: Overall Study
Arm/Group | Experimental: Optimal- 18 Weeks | Experimental: Sub-optimal With AC | Experimental: Optimal With AC | Experimental: Sub-optimal no AC
Started | 27 | 3 | 0 | 2
Completed | 25 | 3 | 0 | 2
Not Completed | 2 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 2 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: No participants received less than 18 weeks (6 cycles) of paclitaxel, carboplatin, trastuzumab and pertuzumab, followed by initiation of doxorubicin and cyclophosphamide.
Groups:
- Total: Total of all reporting groups
Arm/Group | Experimental: Optimal- 18 Weeks | Experimental: Sub-optimal With AC | Experimental: Optimal With AC | Experimental: Sub-optimal no AC | Total
Number analyzed (Participants) | 27 | 3 | 0 | 2 | 32
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 22 | 3 | 0 | 2 | 27
  >=65 years | 5 | 0 | 0 | 0 | 5
Age, Continuous [Median (Full Range); unit: years] | 51 [29 to 81] | 48 [36 to 62] |  | 45 [38 to 54] | 50 [29 to 81]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27 | 3 | 0 | 2 | 32
  Male | 0 | 0 | 0 | 0 | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 27 | 3 |  | 2 | 32

OUTCOME MEASURES:

1. Primary Outcome: Percent of Patients Who Achieve a pCR
Description: pCR is pathologic complete response defined as ypT0/isN0 on pathology report
Time Frame: at surgery post approximately 18 weeks of treatment
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Experimental: Optimal- 18 Weeks | Experimental: Sub-optimal With AC | Experimental: Optimal With AC | Experimental: Sub-optimal no AC
Number analyzed (Participants) | 25 | 3 | 0 | 2
Participants | 19 | 2 | 0 | 0

2. Primary Outcome: Number of of Patients Who Develop Major Toxicities as Defined in Protocol.
Description: Defined based on CTCAE version 4:
  1. Neutropenia (grade>2)
  2. Thrombocytopenia (grade >2)
  3. Anemia (grade >2)
  4. Diarrhea (any grade, grade >3)
  5. Neuropathy (any grade, grade 2, grade >3)
  6. Vomiting (any grade, grade >3)
Time Frame: From start of neo-adjuvant treatment through approximately 18 weeks.
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Experimental: Optimal- 18 Weeks | Experimental: Sub-optimal With AC | Experimental: Optimal With AC | Experimental: Sub-optimal no AC
Number analyzed (Participants) | 25 | 3 | 0 | 2
Participants
  ANC | 19 | 3 |  | 2
  Thrombocytopenia | 2 | 2 |  | 0
  Anemia | 20 | 3 |  | 2
  Diarrhea | 23 | 3 |  | 2
  Neuropathy | 5 | 0 |  | 0
  Vomiting | 5 | 1 |  | 0

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the time a signed and dated ICF is obtained until 3 months post-operative, or until the subject withdrew consent from study participation, whichever occurs first.
Arm/Group | Experimental: Optimal- 18 Weeks | Experimental: Sub-optimal With AC | Experimental: Sub-optimal no AC
All-Cause Mortality (participants affected / at risk) | 1/25 | 0/3 | 0/2
Serious Adverse Events (participants affected / at risk) | 5/25 | 2/3 | 1/2
Other Adverse Events (participants affected / at risk) | 25/25 | 3/3 | 2/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Experimental: Optimal- 18 Weeks (N=25) | Experimental: Sub-optimal With AC (N=3) | Experimental: Sub-optimal no AC (N=2)
Diarrhea (Gastrointestinal disorders) | 1 | 1 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 0 | 0
Back pain (General disorders) | 0 | 0 | 1
Renal calculi (Renal and urinary disorders) | 0 | 0 | 1
Dehydration (General disorders) | 1 | 1 | 0
Enterocolitis (Gastrointestinal disorders) | 0 | 1 | 0
Cellulitis (Infections and infestations) | 0 | 1 | 0
Flank pain (General disorders) | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 0 | 1
Sepsis (Infections and infestations) | 0 | 0 | 1
Anemia (Blood and lymphatic system disorders) | 0 | 0 | 1
Hypokalemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Alanine aminotransferase increased (Investigations) | 0 | 0 | 1
Salmonella infection (Gastrointestinal disorders) | 1 | 0 | 0
Skin infection (Infections and infestations) | 1 | 1 | 0
Kidney infection (Infections and infestations) | 0 | 0 | 1
Typhitis (Gastrointestinal disorders) | 0 | 1 | 0
Neutropenia (Investigations) | 0 | 1 | 0
Breast infection (Infections and infestations) | 1 | 0 | 0
Breast pain (Reproductive system and breast disorders) | 1 | 0 | 0
Progression of disease (General disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Experimental: Optimal- 18 Weeks (N=25) | Experimental: Sub-optimal With AC (N=3) | Experimental: Sub-optimal no AC (N=2)
Neutrophil count increase (Investigations) | 23 | 2 | 2
Thrombocytopenia (Investigations) | 3 | 2 | 1
Anemia (Blood and lymphatic system disorders) | 22 | 2 | 1
Diarrhea (Gastrointestinal disorders) | 23 | 3 | 1
Neuropathy (Nervous system disorders) | 6 | 0 | 0
Vomiting (Gastrointestinal disorders) | 10 | 1 | 1
Alanine aminotransferase increased (Investigations) | 0 | 1 | 0
White blood cell count decreased (Investigations) | 0 | 1 | 0
Hypophosphatemia (Metabolism and nutrition disorders) | 0 | 1 | 1
Hypokalemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Fever (General disorders) | 0 | 0 | 1
Sinus tachycardia (Cardiac disorders) | 0 | 0 | 1
Hypotension (Vascular disorders) | 1 | 0 | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Infusion related reaction (Infections and infestations) | 1 | 0 | 0
Anaphylaxis (Immune system disorders) | 1 | 0 | 0
Upper respiratory infection (Infections and infestations) | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-05-07): https://cdn.clinicaltrials.gov/large-docs/57/NCT02789657/Prot_SAP_000.pdf